CLINICAL TRIAL: NCT04216225
Title: Prospective Observational Multi-center Analysis of Pre-hospital Tourniquet in Extremity Injury
Brief Title: Pre-hospital Tourniquet in Extremity Injury
Status: Enrolling by invitation | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 098.GME.2017.D
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Extremity Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: pre-hospital tourniquet placement — patients with extremity injuries presenting with or without pre-hospital tourniquet placement.

SUMMARY:
2.1. Objective:

• Primary Objective: To compare outcomes of patients with extremity injuries presenting with or without pre-hospital tourniquet placement.

2.2. Study Outcome Measures

* Primary Outcome: Incidence of arrival in shock (SBP <90)
* Secondary Outcomes: Demographics, comorbidities, mechanism of injury, cause of injury, diagnosis codes, procedure codes, Injury Severity Scale, Abbreviated Injury Scale, operative management vs. non-operative management, radiologic findings, pathologic findings, tourniquet effectiveness (as determined both subjectively by trauma surgeon and objectively by presence vs. absence of pulse below level of tourniquet application), total number of units of blood products transfused within first 24 hrs, total number of units of blood products for index admission, type of blood products or other fluid given, hospital length of stay, ICU length of stay, ventilator days, infectious complications, other complications, discharge disposition, 24 hr mortality, overall mortality.

DETAILED DESCRIPTION:
This is a prospective, observational study. All patients who present to the participating ED's who meet inclusion/exclusion criteria will be identified by the treating trauma surgeons. Data collected will include basic patient demographics, data regarding the patient's injuries, data regarding tourniquet use, and data regarding outcomes. Please see the attached data collection tool for specifics (Appendix 12.1). Data will be collected prospectively in an observational manner using the data collection tool. Data collected on individual collection sheets will be de-identified. We plan to complete the data collection and analysis by 01\01\2021.

ELIGIBILITY:
Inclusion Criteria:

≥ 18 y/o Patients with extremity injuries

* With a tourniquet in place OR
* Who the treating physician deems could have benefited from tourniquet placement

Exclusion Criteria:

* Children
* Prisoners
* Pregnant women
* Patients with non-traumatic bleeding requiring tourniquet use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who present to the participating ED's who meet inclusion/exclusion criteria will be identified by the treating trauma surgeons.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of arrival in shock | First 24 hours .
  (Systolic Blood Pressure <90 mmHg (Millimeter of mercury))

CONTACTS AND LOCATIONS:
Overall Officials: Michael Truitt, M.D., Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided